CLINICAL TRIAL: NCT06092437
Title: TAILOR-AHF: Randomized Trial Investigating a Tailored Diuretic Algorithm in Acute Heart Failure Patients
Brief Title: Investigating a Tailored Diuretic Algorithm in Acute Heart Failure Patients
Acronym: TAILOR-AHF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zuyderland Medisch Centrum (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Z2021110
Record Dates: First submitted 2023-08-31; First posted 2023-10-23 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-01

CONDITIONS: Heart Failure Acute
Keywords: Decongestion; Heart failure; Natriuresis; Urinary Sodium
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tailored, Urine sodium guided, intensified diuretic strategy (Experimental)
  Interventions: Other: Urine sodium guided diuretic algorithm
- Usual care (Active Comparator)
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Urine sodium guided diuretic algorithm — Loop diuretics are administered intravenously as soon as possible after diagnosis of ADHF and continued 3dd until recompensation. Spot urine sodium is measured 2 hours after administration of the first in-hospital IV diuretic dose and repeated until the target of 100mmol/L is reached in the first 72 hours of admission (after which, UrNa will be measured once daily). When target is not met, the next dosage of loop diuretic is doubled (max 3dd 250mg furosemide) and thereafter, other diuretics (thiazide, MRA) are added. Acetazolamide in the first 72 hours is advised as background therapy in both treatment arms.
  Arms: Tailored, Urine sodium guided, intensified diuretic strategy
Other: Usual care — Treatment with IV loop diuretics left to the discretion of the treating physician. Acetazolamide in the first 72 hours is advised as background therapy in both treatment arms.
  Arms: Usual care

SUMMARY:
Acutely decompensated heart failure (ADHF) is highly prevalent and has a high (financial) burden on the health care system. Treatment often consists of the administration of IV decongestive agents. Adequate dosing is difficult due to varying diuretic resistance and inadequate parameters to evaluate the response. Urine sodium is a promising biomarker to evaluate the diuretic response. It is hypothesized that a tailored, urine sodium guided diuretic algorithm will result in faster and more complete decongestion and therefore lead to better survival (in terms of mortality and heart failure events) while being non-inferior in terms of safety (mainly regression of kidney function).

DETAILED DESCRIPTION:
Rationale: Acutely decompensated heart failure is a highly prevalent diagnosis with a high burden on resources and a high risk of mortality and re-hospitalization. The prescription of diuretics to relieve congestion has been the cornerstone of treatment for years, but evidence about diuretic response and adequate dosing is still lacking. Inadequate diuretic response (and insufficient decongestion) has a negative influence on outcome but is often not timely addressed. Urinary sodium (Ur-Na) is a promising biomarker in the prediction of diuretic response to the prescribed dose. It is hypothesized that an Ur-Na based, intensified algorithm can help tailor diuretics in an individual way, but sufficient evidence to support its implementation is lacking.

Objective: Investigate if a tailored diuretic algorithm based on Ur-Na has a positive effect on a primary endpoint of reduction in a combined endpoint of death, heart failure events and change in the Kansas City questionnaire total symptom score (KCCQ-TSS) versus standard clinical care in patients hospitalized with AHF, without imposing safety concerns (e.g. worsening renal function).

Study design: Prospective, Single-Blinded, Randomized, Blinded-endpoint trial

Study population: Patients admitted with acutely decompensated heart failure (diagnosed according to the 2021 ESC (European Society of Cardiology) guidelines) who are 18 year or older.

Intervention: Arm I: Tailored, Ur-Na based, intensified diuretic strategy; Arm II: Usual care

Main study parameters/endpoints: Hierarchical composite endpoint of all-cause death, heart failure events and a 4-point or greater difference in Kansas City questionnaire total symptom score (KCCQ-TSS); assessed using a win-ratio approach.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years;
* HF (HFrEF, HFmrEF or HFpEF) diagnosed according to the 2021 HF Guidelines of the European Society of Cardiology [5];
* Presentation with AHF meaning at least one symptom (dyspnea, orthopnea, or edema) and one sign (rales, peripheral edema, ascites, or pulmonary vascular congestion on chest radiography) of AHF;
* An elevated NT-proBNP >300pg/ml;
* Requiring the need for iv diuretics.

Exclusion Criteria:

* Terminal renal insufficiency defined as: dialysis patients or eGFR (estimated glomerular filtration rate) < 10 mL/min/1.73 m2;
* Patients included in other investigational studies regarding heart failure.
* Presentation with cardiogenic shock or respiratory insufficiency or another reason requiring admission to the intensive care unit upon admission (IC transfer later in the hospitalization is not an exclusion).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 466 (Estimated)
Dates: Start 2023-02-27 (Actual); Primary Completion 2026-06-27 (Estimated); Study Completion 2026-08-27 (Estimated)

PRIMARY OUTCOMES:
Hierarchical composite of all-cause mortality, heart failure events and delta quality of life at 90 days follow-up. | 90 days after inclusion
  The primary endpoint is a hierarchical composite calculated using a win-ratio approach of:
  i) Mortality (all-cause) at 90 days after hospitalization; ii) Heart failure events at 90 days after hospitalization (1. a >2 times increase in oral loop diuretic dose, 2. the need for iv administration of loop diuretics, 3. an emergency department visit or hospitalization for HF), wherein a single event or hospitalization will be sufficient to reach the combined endpoint; iii) Delta in quality of life measured using the Kansas City Cardiomyopathy Questionnaire total symptom score (KCCQ-TSS) from baseline to 90 days after hospitalization

SECONDARY OUTCOMES:
Delta NT-pro BNP | From admission to discharge and 90 days after hospitalisation
  Delta NT-proBNP from admission to discharge and 90-days follow up
Successful decongestion | Day 3 after inclusion
  Number of participants with successful decongestion (defined as a clinical congestion score of 2 or less and NYHA I-II)
Change in clinical congestion score | From date of randomization until date of hospital discharge (regarding initial hospitalisation at time of randomisation, assessed up to 90 days),
  Change in clinical congestion score from admission to discharge
Quality of life (Kansas City Cardiomyopathy Questionnaire) | 90 days after inclusion
  Quality of life assessed using the Kansas City Cardiomyopathy Questionnaire
Adverse (safety) events | 90 days after inclusion
  All-cause readmissions at 90-days, all-cause and cardiovascular mortality at 90-days, (symptomatic) hypotension, hypokalemia, urinary tract infection, phlebitis, atrial fibrillation, fall/trauma and decompensated HF
All-cause mortality and heart failure readmissions | 14 days after inclusion
  All-cause mortality and heart failure readmissions at 14 days follow up
All-cause mortality and heart failure readmissions | 6 months after inclusion
  All-cause mortality and heart failure readmissions at 6 months follow up
Chronic dialysis | 90 days after inclusion
  Occurence of the need for chronic dialysis at 90-days follow up
Days alive outside the hospital | 90 days after inclusion
  Days alive outside the hospital at 90-days follow up
Time to first heart failure hospitalization and number of heart failure hospitalizations | 90 days after inclusion
  Time to first heart failure hospitalization and number of heart failure hospitalizations
Number of outpatient visits | 90 days after inclusion
  Number of outpatient visits in the first 90 days
Number of worsening heart failure events | 90 days after inclusion
  Number of worsening heart failure events at 90 days:
  i) a >2 times increase in oral loop diuretic dose, ii) the need for iv administration of loop diuretics, iii) an emergency department visit or hospitalization for HF
Delta weight | From date of randomization until date of hospital discharge (regarding initial hospitalisation at time of randomisation, assessed up to 90 days)
  Delta weight (in kilograms) from admission to discharge
Hospital length of stay | Number of days from hospitalization untill end of clinical treatment (not including days waiting for post-hospital care) or hospital discharge, whichever came first, assessed up to 90 days after randomization.
  Number of days from hospitalization untill discharge or end of clinical treatment (not including days waiting for post-hospital care)
Worsening renal function | Baseline until 90 days follow-up
  Delta creatinine from baseline until discharge and 90 days follow-up

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - Zuyderland MC, Heerlen, Limburg
  - Amphia ziekenhuis, Breda, North Brabant

IPD SHARING:
Plan to Share IPD: No